CLINICAL TRIAL: NCT05564637
Title: Comprehensive O2 Transfer Analysis From the Lung to Mitochondria of Inhaled Treprostinil in Interstitial Lung Disease Pulmonary Hypertension
Brief Title: A Study of Treprostinil to Treat Interstitial Lung Disease Pulmonary Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: United Therapeutics (Industry)
Responsible Party: Principal Investigator, Yogesh Reddy, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-004971
Record Dates: First submitted 2022-09-28; First posted 2022-10-03 (Actual); Results first posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Pulmonary Arterial Hypertension; Interstitial Lung Disease; Healthy Adults
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Lung Diseases, Interstitial | interventions — treprostinil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Healthy Volunteers (Other): Healthy volunteers will undergo RHC while exercising and an optional muscle biopsy.
  Interventions: Diagnostic Test: Right Heart Catheterization (RHC) while exercising; Diagnostic Test: Optional Muscle Biopsy
- PAH-ILD Patients (Experimental): Patients diagnosed with PAH-ILD will undergo RHC while exercising, receive inhaled treprostinil, and undergo an optional muscle biopsy.
  Interventions: Drug: Treprostinil; Diagnostic Test: Right Heart Catheterization (RHC) while exercising; Diagnostic Test: Optional Muscle Biopsy

INTERVENTIONS:
Drug: Treprostinil — 30mcg (5 breaths) of inhaled treprostinil will be administered during the RHC procedure and patients will be initiated on outpatient inhaled treprostinil therapy for 3-months with gradual up titration to target dose as per standard clinical practice.
  Arms: PAH-ILD Patients
Diagnostic Test: Right Heart Catheterization (RHC) while exercising — A procedure to measure how well or poorly your heart is pumping and to measure the pressures in the heart and lungs. A catheter will be inserted into a vein and artery in order to take the measurements and this will be conducted while exercising on a supine cycle ergometer. Various measurements will be taken during periods of rest and exercise.
Diagnostic Test: Optional Muscle Biopsy — A sample of muscle tissue will be collected and analyzed for the ability of the cells to utilize oxygen.

SUMMARY:
The purpose of this research study is to find out more about the drug treprostinil via inhaler and the mechanisms of why patients with pulmonary arterial hypertension related to Interstitial Lung disease (PAH-ILD) have limitations during exercise. The investigator is studying treprostinil's effect on patients with PAH-ILD during exercise and its effect on their quality of life after using it for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Pulmonary Arterial Hypertension due to Interstitial Lung Disease (ILD-PAH) being considered for inhaled treprostinil
* Resting right heart catheterization with mean pulmonary artery pressure >20 mmHg and PVR> 3 Wood units
* Healthy volunteers will have no known lung disease, heart failure, muscular disease or pulmonary hypertension, no bleeding abnormalities, and have the ability to exercise.

Exclusion Criteria:

* Inability to exercise
* Females who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2023-03-13 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yogesh N Reddy, M.B.B.S, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 29 subjects were consented of which 5 screen failed prior to study group assignment.
Period: Overall Study
Arm/Group | Healthy Volunteers | PAH-ILD Patients
Started | 1 | 23
Completed | 1 | 22
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Population: Only 1 participant was enrolled in the healthy volunteers arm. Based on the low enrollment number in the healthy volunteers arm, no data is reported for the 1 subject in order to protect and maintain participant privacy/confidentiality.
Groups:
- PAH-ILD Patients: Patients diagnosed with PAH-ILD underwent RHC while exercising, received inhaled treprostinil, and underwent an optional muscle biopsy.
  Treprostinil: 30mcg (5 breaths) of inhaled treprostinil was administered during the RHC procedure and patients were initiated on outpatient inhaled treprostinil therapy for 3-months with gradual up titration to target dose as per standard clinical practice.
  Right Heart Catheterization (RHC) while exercising: A procedure to measure how well or poorly your heart is pumping and to measure the pressures in the heart and lungs. A catheter was inserted into a vein and artery in order to take the measurements and this was conducted while exercising on a supine cycle ergometer. Various measurements were taken during periods of rest and exercise.
  Optional Muscle Biopsy: A sample of muscle tissue were collected and analyzed for the ability of the cells to utilize oxygen.
- Healthy Volunteers: Healthy volunteers underwent RHC while exercising and an optional muscle biopsy.
- Total: Total of all reporting groups
Arm/Group | PAH-ILD Patients | Healthy Volunteers | Total
Number analyzed (Participants) | 23 | 0 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.5 (8) |  | 72.5 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 0 | 10
  Male | 13 | 0 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 18 | 0 | 18
  Unknown or Not Reported | 5 | 0 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 17 | 0 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 0 | 5
Region of Enrollment [Number; unit: participants]
  United States | 23 |  | 23

OUTCOME MEASURES:

1. Primary Outcome: Cardiac Output Reserve (Qc)
Description: Cardiac output reserve (Qc) is the difference between the heart's maximum output during exercise and its resting output. This was measured using the direct Fick method (L/min).
Time Frame: Baseline, approximately 35 minutes
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Liters/Min
Arm/Group | PAH-ILD Patients | Healthy Volunteers
Number analyzed (Participants) | 22 | 0
Liters/Min
  Baseline | 3.3 (2.1) |
  Approximately 35 minutes | 3.8 (1.8) |

2. Secondary Outcome: Ventilatory Efficiency (VE/VCO2)
Description: Ventilatory efficiency was assessed as a ratio between the ventilation (VE) and carbon dioxide production (VCO2) measured during the RHC procedure. VE/VCO2 evaluates how efficiently a person breathes during exercise.
Time Frame: Baseline, approximately 35 minutes
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | PAH-ILD Patients | Healthy Volunteers
Number analyzed (Participants) | 16 | 0
Ratio
  Baseline | 50.4 (10.6) |
  Approximately 35 Minutes | 51.2 (11.2) |

3. Secondary Outcome: New York Heart Association (NYHA) Functional Class
Description: Participants severity of heart failure symptoms was classified according to the NHYA functional class (I-IV). Lower classifications indicate lower severity of heart failure symptoms.
Time Frame: Baseline, 3-months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | PAH-ILD Patients | Healthy Volunteers
Number analyzed (Participants) | 22 | 0
Participants
  NYHA I | 1 |
  NYHA II | 9 |
  NYHA III | 6 |
  NYHA IV | 6 |

4. Secondary Outcome: Resting Pulmonary Vascular Resistance
Description: Resting pulmonary vascular resistance was measured in Wood units (mm Hg/L/min) during the RHC procedure. Resting pulmonary vascular resistance is the resistance against blood flow from the pulmonary veins to the left atrium of the heart.
Time Frame: Baseline; after 30 minutes of rest
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mm Hg/L/min
Arm/Group | PAH-ILD Patients | Healthy Volunteers
Number analyzed (Participants) | 22 | 0
mm Hg/L/min
  Baseline | 5.4 (2.1) |
  After 30 minutes of Rest | 3.1 (1.4) |

5. Secondary Outcome: Exercise Pulmonary Vascular Resistance
Description: Exercise pulmonary vascular resistance was measured in Wood units (mm Hg/L/min) during the RHC procedure.
Time Frame: Baseline; approximately 35 minutes
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mm Hg/L/min
Arm/Group | PAH-ILD Patients | Healthy Volunteers
Number analyzed (Participants) | 22 | 0
mm Hg/L/min
  Baseline | 4.3 (2.1) |
  Approximately 35 minutes | 2.2 (1.2) |

6. Secondary Outcome: Resting Pulmonary Artery Pressure
Description: Resting pulmonary artery pressure (mmHg) was measured during the RHC procedure. Pulmonary artery pressure is the pressure within the pulmonary arteries, which transport deoxygenated blood from the right side of the heart to the lungs for oxygenation.
Time Frame: Baseline; after 30 minutes of rest
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | PAH-ILD Patients | Healthy Volunteers
Number analyzed (Participants) | 22 | 0
mmHg
  Baseline | 36.0 (7.3) |
  After 30 minutes of Rest | 25.1 (5.2) |

7. Secondary Outcome: Exercise Pulmonary Artery Pressure
Description: Exercise Pulmonary artery pressure (mmHg) was measured during the RHC procedure. Pulmonary artery pressure is the pressure within the pulmonary arteries, which transport deoxygenated blood from the right side of the heart to the lungs for oxygenation.
Time Frame: Baseline; approximately 35 minutes
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | PAH-ILD Patients | Healthy Volunteers
Number analyzed (Participants) | 22 | 0
mmHg
  Baseline | 50.4 (9.3) |
  Approximately 35 Minutes | 40.6 (9.0) |

8. Secondary Outcome: Resting Right Atrial Pressure
Description: Resting right atrial pressure (mmHg) was measured during the RHC procedure. Right atrial pressure is a measurement that reflects the amount of blood returning to the heart and the heart's ability to pump blood into the arterial system.
Time Frame: Baseline; after 30 minutes of rest
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | PAH-ILD Patients | Healthy Volunteers
Number analyzed (Participants) | 22 | 0
mmHg
  Baseline | 7.9 (3.4) |
  After 30 Minutes of Rest | 6.2 (3.1) |

9. Secondary Outcome: Exercise Right Atrial Pressure
Description: Exercise right atrial pressure (mmHg) was measured during the RHC procedure. Right atrial pressure is a measurement that reflects the amount of blood returning to the heart and the heart's ability to pump blood into the arterial system.
Time Frame: Baseline; approximately 35 minutes
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | PAH-ILD Patients | Healthy Volunteers
Number analyzed (Participants) | 22 | 0
mmHg
  Baseline | 16.1 (6.3) |
  Approximately 35 Minutes | 12.9 (6.0) |

ADVERSE EVENTS:
Time Frame: Major procedural complications were collected from the time of informed consent through study completion, approximately 4 months.
Description: Adverse event definition used in this study: Major procedural complications were reported through the data collection form and were monitored and adjudicated by the PI. Adverse events were not separately reported to the IRB. The drug inhaled treprostinil represents standard of care therapy for PAH-ILD and the acute administration should post no additional risk compared to the chronic therapy that was subsequently administered at an even higher dose.
Groups:
- Healthy Volunteers: Healthy volunteers underwent RHC while exercising and an optional muscle biopsy.
  Right Heart Catheterization (RHC) while exercising: A procedure to measure how well or poorly your heart is pumping and to measure the pressures in the heart and lungs. A catheter was inserted into a vein and artery in order to take the measurements and this was conducted while exercising on a supine cycle ergometer. Various measurements were taken during periods of rest and exercise.
  Optional Muscle Biopsy: A sample of muscle tissue was collected and analyzed for the ability of the cells to utilize oxygen.
Arm/Group | Healthy Volunteers | PAH-ILD Patients
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/23
Other Adverse Events (participants affected / at risk) | 0/1 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-09): https://cdn.clinicaltrials.gov/large-docs/37/NCT05564637/Prot_SAP_000.pdf